CLINICAL TRIAL: NCT01468415
Title: Efficiency Comparison Between Methylprednisolone and Phenol 8% Treatment Using a Trans Sacral Approach - on Lower Back Pain and Limbs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 58/11
Record Dates: First submitted 2011-11-06; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-05

CONDITIONS: Back Pain
Keywords: Methylprednisolone; trans sacral block; phenol
MeSH Terms: conditions — Back Pain | interventions — Phenol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: phenol — 1 cc of 8% phenol dissolved in water or 20cc of 8o mg Methylprednisolone diluted in 0.25% marcaine.

SUMMARY:
The American Society of Anesthesiologists Task Force on Management, Chronic Pain section, recommended Phenol neurolysis when other techniques have failed to provide adequate pain control. In this study we sought to Compare the pain relieve on a Lower Back and Limbs obtained from Methylprednisolone and Phenol 8% Treatment given by Trans Sacral Approach. The study includes patients who suffers from a chronic low back and/or limbs pain which were referred to be given epidural as a treatment. Control group receives 80 mg Methylprednisolone while the test group receives phenol 8%.

ELIGIBILITY:
Inclusion Criteria: -at least 18 years of age;

* chronic low back pain of at least 12 weeks duration;
* patients which were diagnosed as a candidate for epidural since other techniques have failed to provide adequate pain control
* Sciatica due to Lumbar Disc Herniation
* Neurogenic Claudication due to Lumbar Spinal Stenosis

Exclusion Criteria:

* patients with unbalanced high blood pressure
* patients who can not ley prone
* patients who consumes anti-clotting medications
* patients with bleeding problems
* patients with Diabetes
* patients who suffers from chronic non-specific lower back and limb pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel